CLINICAL TRIAL: NCT02623569
Title: Evaluation of the Anti-anginal Efficacy and Safety of Ivabradine Used in Patients With Stable Effort Angina Pectoris. A 12 Weeks Randomised, Double-blind Controlled, Parallel-group, Multicentre Study
Brief Title: To Assess the Anti-anginal Safety and Efficacy of Ivabradine in Subjects With Stable，Symptomatic Chronic Angina
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xintong Pharmacy Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A130901CSPF01
Record Dates: First submitted 2015-11-29; First posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Angina Pectoris
MeSH Terms: conditions — Angina Pectoris | interventions — Ivabradine; Atenolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivabradine (Experimental): Ivabradine 5 mg twice a day for first 4 weeks and 7.5mg twice a day when positive ETT and HR（heard rate）>60times/min or negative ETT and HR（heard rate）>80times/min of subjects.
  Interventions: Drug: Ivabradine
- Atenolol (Active Comparator): Atenolol 12.5 mg twice a day for first 4 weeks and 25mg twice a day when positive ETT and HR（heard rate）>60times/min or negative ETT and HR （heard rate）>80times/min of subjects.
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Ivabradine — Not Provided
  Other Names: Not Provided
  Arms: Ivabradine
Drug: Atenolol — Not Provided
  Other Names: Not Provided
  Arms: Atenolol

SUMMARY:
Arms Assigned Interventions

Experimental: Ivabradine Ivabradine 5 mg twice a day for first 4 weeks and 7.5mg twice a day when positive ETT and HR>60times/min or negative ETT and HR>80times/min of subjects.

Active Comparator: Atenolol Atenolol 12.5 mg twice a day for first 4 weeks and 25mg twice a day when positive ETT and heard rate>60times/min or negative ETT and HR >80times/min of subjects.

DETAILED DESCRIPTION:
1. Washout period：Chronic angina patients stop using medicine that affect heart rate. The patients undergoes ETT after 2-7 days and positive ETT into the treatment period(If not take similar medicine, patients can be carried out ETT directly)。
2. Treatment period：Patients carried out ETT after therapy with Ivabradine(5mg,bid)/ Atenolol(12.5mg,bid) for 4 weeks.The dose adjust base on test result and heart rate, Ivabradine(5mg,bid)/Atenolol(12.5mg,bid) or Ivabradine(7.5mg,bid)/ Atenolol(25mg,bid) for 8 weeks and carried out ETT.
3. security period：After the treatment period, all patients to take Atenolol 12.5mg/ 25mg bid 1 week.

If heart rate are low 50 times/min after taking Ivabradine 5mg/ Atenolol 12.5mg, subjects should withdrawal and dropped out study. If subjects heart rate are low 50 times/min after taking Ivabradine 7.5mg/ Atenolol 25mg, subjects should change the dose to Ivabradine 5mg/ Atenolol 12.5mg.

ELIGIBILITY:
Inclusion Criteria:

1. male or female aged 18 to 75 years
2. Clearly understand the study and participate in it voluntarily; the informed consent should be signed in person or by legal guardian.
3. Chronic Stable Angina was confirmed by clinic over 3 months.
4. Patients with clinical diagnosis of chronic stable angina and must meet one of the following conditions:

   * Patients who have a history of myocardial infarction over 3 months.
   * Patients who have received coronary intervention or CABG（Coronary Artery Bypass Grafting） over 6 months.
   * Stenosis of more than 50% in at least one major epicardial coronary artery shown by Coronary Angiograph.
   * Ischemic electrocardiogram changes：ST-segment depression ≥ 1.0 mm compared with P-R or elevate≥1.0 mm during exercise ECG Computed Tomography Angiography (CTA) showed more than 50% stenosis with typical angina symptoms
5. ultrasonic cardiogram disclosed that left ventricular ejection fraction ≥50 %.
6. Patients who manifested positive ETT (exercise tolerance testing) (defined as ST-segment depression ≥ 1 mm compared with at rest, with or without limiting angina) at screening.

Exclusion Criteria:

1. Clinically significant Valvular disease, congenital heart disease, pulmonary hypertension, cerebral apoplexy, dissecting aneurysm, hypertrophic cardiomyopathy, acute myocarditis/cp.
2. Patients with myocardial infarction within the preceding 3 months
3. Patients have received Coronary angioplasty or CABG within the preceding 6 months.
4. Patients who have severity vessels disease with left main coronary artery but have no valid treatment.
5. Patients with congestive heart failure(New York Heart Association class III or IV)or acute pulmonary edema.
6. Patients whose rest heart rate< 60 bpm.
7. Patients with nonrespiratory sinus arrhythmia or arrhythmia(e.g.,AVB(auriculo-ventricular block)ⅡⅢ,atrial fibrillation,atrial flutter,SSS(sick sinus syndrome)) or implantable cardiac defibrillator (ICD).
8. Patient with any conditions that interfered the performance of exercise tolerance test or a history of an abnormal exercise response limited by electrocardiograph (ECG) changes.
9. Patient with uncontrolled hypertension (seated systolic blood pressure (SBP）≥180 mmHg or diastolic blood pressure (DBP) ≥100 mmHg); SBP<90 mmHg and/or DBP<60 mmHg
10. Diabetic with uncontrolled blood glucose(FBG≥11.1 mmol/L and/or RBG≥13.6 mmol/L）
11. Patients with anemia(male:Hb≤120 g/L；female：Hb≤110 g/L)
12. Patients complicated with systemic diseases included thyroid dysfunction、glaucoma、cataract，neurological、mental、psychological disease and any other disease that influence the judgment.
13. Severe concurrent pathology, including terminal illness (cancer, AIDS, etc.).
14. Patients with mental or legal disorder.
15. Patients who were suspected addicted into alcohol or drug abuse or with severe complications that would make the condition more complicated assessed by the investigator.
16. People have liver or renal dysfunction (ALT≥2×ULN、AST≥2×ULN、eGFR≤60ml/min/1.73m2）
17. Patients who should use unapproved drug during the study.
18. Patients who accepted amiodarone(in recent 3 months)and/or benzetimide、βblockers（in recent 7 days)、
19. Patients with history of allergy or suspected allergic to the drug（e.g.，Hydrochloric ivabradine,atenolol, βblockers）or lactose.
20. Woman who disagree with contraception during treatment period ，with pregnancy, lactation or positive result of pregnancy test.
21. Patients with Chronic Obstructive Pulmonary Disease (COPD) requiring bronchodilators.
22. Patients who is participating in other trials or has been participated in other trials in recent 3 months
23. Patients who were unable to participate in the study as judged by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is Change from total exercise duration in exercise tolerance test (ETT) | Baseline and end of treatment (Week 12) .

SECONDARY OUTCOMES:
Time to angina in exercise tolerance test. | 12 weeks
Time to 1 mm ST-segment depression in exercise tolerance test | 12 weeks
Number of angina attacks in exercise tolerance test per week | 12 weeks
Number of sublingual nitroglycerin consumption per week | 12 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The General Hospital of Shenyang Military, Shenyang, Liaoning